CLINICAL TRIAL: NCT03957005
Title: A Cardiovascular Risk Assessment Model According to Behavioral, Psychosocial and Traditional Factors in Patients With Myocardial Infarction: A Multi-center Cohort Study
Brief Title: Cardiovascular Risk Assessment Model in Patients With MI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Collaborators: National Institute for Medical Research Development (Unknown)
Responsible Party: Principal Investigator, Masoumeh Sadeghi, Head of Cardiac Rehabilitation Research Center, Isfahan University of Medical Sciences
Other Study IDs: 964708
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Myocardial Infarction, Acute
Keywords: Myocardial Infarction; Major cardiovascular events; Risk assessment
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate life-style and psycho social factors of major cardiovascular events in patients with myocardial infarction in three different provinces of Iran and to design a risk assessment chart for major cardiovascular events in patients with MI.

DETAILED DESCRIPTION:
Patients with pre-existing MI are at higher risk of major cardiovascular events (MCE). Current studies mainly focus on cardiovascular disease (CVD) risk assessment in general population without a history of CVD. Because of high prevalence of ischemic heart disease, especially in developing countries such as Iran, this group of patients form a large high-risk population. Factors such as life styles, habits, and psychosocial features are adjustable factors which have been less studied in relation to MCE in MI patients worldwide. Psychological factors are especially most important in patients with a pre-existing CVD and can account for worse outcomes independent of other pathological factors. The cardiovascular events are multifactorial and control of traditional risk factors such as hypertension and hyperlipidemia cannot efficiently reduce MCE. Identification and comprehensive assessment of MCE risk factors is essential for reducing MCE and thus better management of patients. The effect of different factors on MCE could be analysed using risk assessment model. To the best of our knowledge, this is the first comprehensive study of life style and psychological risk factors in CVD patients and the first time to perform MCE risk assessment modelling in MI patients.

The predictors recorded in this study are categorized in three main issues: 1) lifestyle, including: nutritional status, physical activity, tobacco smoking and drug abuse, sleep quality, and sexual function assessed by relevant questionnaires. 2) behavioral and psychological factors, including: depression, psychological distress, health anxiety, health related quality of life, type D personality, coping strategies, sense of coherence and medication adherence also measured by appropriate questionnaires. 3) Traditional risk factors, including: hypertension, diabetes, and hyperlipidemia which will be extracted from medical and laboratory records of patients and questionnaires. All predictor variables will be assessed in every year follow-up for three years during the study.

ELIGIBILITY:
Inclusion Criteria:

* clinically verified diagnosis of the first episode ST-elevation myocardial infarction
* providing written informed consent

Exclusion Criteria:

* history of prior documented CVD
* living in a nursing home or other institutions
* having a serious medical condition with a survival of less than 3 years
* participation in another scientific study
* not willing to participate in each phase of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will perform in three referral hospitals of Tehran, Isfahan and Bandarabbas counties. Participants of this study will be those hospitalized because of their first myocardial infarction.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-11-06 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of MCE within follow up period | From enrollment up to 36 months of followup
  MCE includes two type of CV events: coronary artery disease-specific (MI, unstable angina (hospitalized angina), coronary revascularization or death from coronary heart disease) and cerebrovascular disease-specific events (ischemic or hemorrhagic stroke, transient ischemic attack, cerebrovascular disease-specific revascularization or death from cerebrovascular disease).

CONTACTS AND LOCATIONS:
Overall Officials: Masoumeh Sadeghi, MD, Principal Investigator — Cardiac Rehabilitation Research Center
Locations (4):
- Iran (4):
  - Dr Heshmat Hospital, Rasht, Gilan Province
  - Shahid Mohammadi hospital, Bandar Abbas, Hormozgan
  - Chamran Cardiology Hospital, Isfahan
  - Shahid Rajaei hospital, Tehran

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after study publication.